CLINICAL TRIAL: NCT04463602
Title: A Phase 2b, Multicenter, Open-label, Randomized, Comparator-Controlled, Study to Evaluate the Efficacy and Safety of Desidustat Tablet for the Management of COVID-19 Patients
Brief Title: Desidustat in the Management of COVID-19 Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DESI.20.004
Record Dates: First submitted 2020-07-07; First posted 2020-07-09 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — desidustat; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Desidustat + Standard of Care (Experimental): Test: Desidustat + Standard of care
  Desidustat 100 mg for the duration of 14 days along with the recommended standard of care at the time of conduct of trial.
  Interventions: Drug: Desidustat; Other: Standard of Care
- Standard of Care (Active Comparator): Control: Standard of care
  Standard of care treatment for the duration of 14 days at the time of conduct of trial.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Desidustat — 100 mg once daily
  Arms: Desidustat + Standard of Care
Other: Standard of Care — Standard of care as per local authority

SUMMARY:
This study is a Phase 2b, Multicenter, Open-label, Randomized, Comparator- Controlled Study to Evaluate the Efficacy and Safety of Desidustat Tablet for the Management of mild, moderate and severe COVID-19 patients. 100 mg of Desidustat will be administered for a period of 14 days along with recommended standard care during the trial.

DETAILED DESCRIPTION:
This is a phase 2b, multicenter, open-label, randomized, comparator-controlled clinical trial to evaluate the efficacy and safety of Desidustat for the management of COVID-19 patients. First 12 mild to moderate subjects (Test arm: Desidustat + Standard of care arm, 06 subjects and Reference arm: Standard of care, 06 subjects) will be enrolled in the study and after evaluation of safety of these 12 subjects by Data Monitoring Committee other 12 severe subjects (Test arm: Desidustat + Standard of care arm, 06 subjects and Reference arm: Standard of care arm, 06 subjects) will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to comprehend and willingness to sign a written ICF by the subject/impartial witness.
2. Male and Females, age ≥18 years at enrollment.
3. Understands and agrees to comply with planned study procedures.
4. Agrees to the collection of pharyngeal swabs and blood sample as per protocol.
5. Has laboratory-confirmed SARS-CoV-2 infection as determined by PCR, or other commercial or public health assay in any specimen within one week.
6. Illness of any duration, and at least one of the following:

   1. Radiographic infiltrates by imaging (chest x-ray)
   2. Clinical assessment (evidence of rales/crackles or other clinical symptoms on exam).
7. Women of childbearing potential must agree to use at least one primary form of contraception for the duration of the study (acceptable methods will be determined by the site).

Exclusion Criteria:

1. ALT/AST >5 times the upper limit of normal.
2. Stage V CKD (i.e. eGFR <15 ml/min/1.73 m2 or requiring dialysis).
3. Pregnant or breast feeding.
4. Severe co-morbidity (e.g. uncontrolled hypertension and uncontrolled DM, systemic disease which affect the vital organs severity, immunocompromised patients etc.) as per investigator's assessment.
5. Comorbid condition like myocardial infarction or heart failure within 90 days of recruitment.
6. Prolong QT interval (>450 ms).
7. Patients on invasive mechanical ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2020-07-25 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Clinical status of subject on a 7-point ordinal scale | Week 2
  1. Not hospitalized, no limitations on activities.
  2. Not hospitalized, limitation on activities.
  3. Hospitalized, not requiring supplemental oxygen.
  4. Hospitalized, requiring supplemental oxygen.
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices.
  6. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO).
  7. Death.

SECONDARY OUTCOMES:
PCR test | Week 2 and Week 4
  PCR for SARS-CoV-2 in pharyngeal swab
Supplemental Oxygen | Week 2 and Week 4
  Occurrence of supplemental Oxygen
Mechanical Ventilation | Week 2 and Week 4
  Occurrence of Mechanical Ventilation
Incidence of Treatment-Emergent Adverse Events | Week 2 and Week 4
  Occurence of Adverse events
Laboratory Assessments | Week 2 and Week 4
  Laboratory Assessments
C-reactive protein (CRP) | Week 2 and Week 4
  Inflammatory Biomarker
Interleukin 6 (IL-6) | Week 2 and Week 4
  Inflammatory Biomarker
D-dimer | Week 2 and Week 4
  Inflammatory Biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Dr Deven Parmar, MD, Study Director — Cadila Healthcare Ltd.
Locations (1):
- Avant Sante Site 1, Monterrey, Mexico

IPD SHARING:
Plan to Share IPD: No